CLINICAL TRIAL: NCT05558384
Title: The Influence of Excess Adiposity on Cardiorespiratory, Insulin-like Growth Factor, and Metabolic Responses to a Standardized Aerobic Exercise Program in Cancer Survivors
Brief Title: Influence of Adiposity on IGF-1 and Fitness Response to Exercise in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0356.ccc
Record Dates: First submitted 2022-09-19; First posted 2022-09-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Overweight and Obesity
MeSH Terms: conditions — Neoplasms; Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single-arm feasibility pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic exercise (Experimental): 15-week standardized aerobic exercise intervention
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — A 15-week standardized aerobic exercise intervention.
  * Frequency: 5 days/wk (2 supervised)
  * Intensity: 50-59% heart rate reserve
  * Time: 40 min/session (ramp up from 25-40 during first 4 weeks)
  * Type: Aerobic exercise (e.g. treadmill, walking/jogging, cycling, elliptical)

SUMMARY:
This is a pilot feasibility study of an investigation of the influence of excess adiposity on cardiorespiratory fitness (CRF), insulin-like growth factor-1 (IGF-1), and metabolic responses to a standardized aerobic exercise program in cancer survivors. This investigation attempts to isolate the influence of adiposity on these responses. We will enroll overweight, obese, and normal weight cancer survivors with a primary diagnosis of breast, prostate, or colorectal cancer who have completed all cancer-related treatment. Participants will engage in a 15-week aerobic exercise intervention with pre- and post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* Primary cancer diagnosis of breast, prostate, or colorectal cancer
* Completion of all cancer-related treatment > than 6 months prior and < 5 years prior to enrollment
* Ability and willingness to participate in a supervised exercise program

  * All participants will be required to obtain a signed physician clearance to participate in exercise form prior to enrollment

Exclusion Criteria:

* Presence of a secondary active cancer diagnosis or metastatic disease
* Any current cancer treatment (including hormonal treatment) or planned cancer treatment in the next 5 months
* Greater than 100 min of self-reported regular exercise per week
* BMI < 18.5 (underweight)
* Any significant metabolic condition, such as diabetes. Individuals with pre-diabetes or metabolic syndrome will not be excluded, but this information will be recorded.
* Any medical condition that would impact the safety of, or participation in, an exercise program or exercise testing, including:

  * Orthopedic conditions such as advanced osteoarthritis, mobility-limiting amputations or chronic injuries, or mobility-limiting acute orthopedic injuries
  * Advanced rheumatoid arthritis or chronic widespread pain conditions such as fibromyalgia
  * Pulmonary conditions such as chronic obstructive pulmonary disease, emphysema, or interstitial lung disease
  * Known cardiovascular disease, uncontrolled hypertension, or new cardiac event within the past 6 months

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | up to 12 months
  Number of participants joining the study per month
Study Adherence | up to 12 months
  Percentage of participants completing pre- and post-intervention assessments
Intervention Adherence | 15 weeks
  Average percentage of prescribed exercise sessions completed by participants

SECONDARY OUTCOMES:
Serum IGF-1 | Baseline, Week 15
  Collected via venipuncture
Estimated VO2max | Baseline, Week 15
  Maximal oxygen consumption estimated from a 3 minute step test (Tecumseh Step Test)
Total visceral adiposity | Baseline, Week 15
  Collected with dual-energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Marker, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot feasibility investigation. Data may be made available upon request. Future, fully powered investigations with include an IPD.